CLINICAL TRIAL: NCT02805816
Title: Choosing a Preferred Serology Kit for Screening and Diagnosis of Celiac Disease
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, raanan shamir, Prof, Rabin Medical Center
Other Study IDs: 0466-15 RMC
Record Dates: First submitted 2016-06-08; First posted 2016-06-20 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Tissue transglutaminase; Histology
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10 cc of blood samples (for celiac serology kits assessment)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: Children with suspicion of CD based on positive serology (TG2 >2 times upper limit of normal) and classical clinical manifestations or belonging to high risk groups, who underwent gastroscopy with intestinal biopsies.
- Control group: Children without suspicion of CD who underwent gastroscopy and duodenal biopsies for other reasons (abdominal pain, failure to thrive, vomiting, eg)

SUMMARY:
The investigators will perform prospective observational multicenter study which includes children with suspicion of CD who referred to gastroscopy and intestinal biopsies (study group) and children without suspicion of CD who underwent gastroscopy for other reasons. The investigators will compare sensitivity, specificity and predictive values of several serological kits of TG2 (tissue transglutaminase) (Bioplex 2200, Bioflash, Phadia 250, Liason-XL, Orgentec Alergia and Eurospital) compared with definitive diagnosis of CD according to histological findings.

DETAILED DESCRIPTION:
Small bowel biopsies have so far been considered as the reference standard for the diagnosis of Celiac disease (CD). However, during the last decades evidence has accumulated on the diagnostic value of specific CD antibodies and has increasingly been used for diagnostic purposes. At the same time, the leading role of histology for the diagnosis of CD has been questioned for several reasons: histological findings are not specific for CD, lesions may be patchy and can occur in the duodenal bulb only and interpretation depends on preparation of the tissue and is prone to a high inter-observer variability. The diagnosis of CD may then depend not only on the results of small bowel biopsies, but also on information from clinical data and on results from specific CD antibody testing. ESPGHAN (European Society of Gastroenterology, Hepatology and Nutrition) guidelines for the diagnosis of CD which was recently published enabled diagnosis of CD based on classical symptoms and high titre levels (>10 times upper limit of normal) of tissue transglutaminase (TG2) and positive Endomysial Anti bodies (EMA) in separate blood samples.

Due to these facts, it is important to use serological kit for TG2 with high specificity and sensitivity. The aim of this study is to assess in a prospective study the kit with the highest sensitivity and specificity among patients with suspected CD.

The investigators will perform prospective observational multicenter study which includes children with suspicion of CD who referred to gastroscopy and intestinal biopsies (study group) and children without suspicion of CD who underwent gastroscopy for other reasons. The investigators will compare sensitivity, specificity and predictive values of several serological kits of TG2 (Bioplex 2200, Bioflash, Phadia 250, Liason-XL, Orgentec Alergia and Eurospital) compared with definitive diagnosis of CD according to histological findings.

ELIGIBILITY:
Inclusion Criteria:

1. Child with clinical suspicion of CD (chronic or recurrent diarrhea, Failure to thrive, growth impairment , iron deficiency anemia, vomiting, chronic abdominal pain, abdominal distension , constipation, fatigue, recurrent oral aphthous or dermatitis herpetiformis) and high TG2 serology (>2 times upper limit of normal) who is referred to gastroscopy and intestinal biopsies Or
2. Asymptomatic child who belongs to high risk group of celiac (Diabetes mellitus type 1, Hashimoto thyroiditis, Down syndrome, Turner syndrome, Williams syndrome, Auto-immune Hepatitis or first degree with CD) and high TG2 serology (>2 times upper limit of normal) who is referred to gastroscopy and intestinal biopsies .

   and
3. signed consent form

Exclusion Criteria:

1. IgA (Immunoglobulin A) deficiency
2. Malignancy
3. Inflammatory Bowel Disease
4. Severe chronic infection (HIV, Tuberculosis)
5. Primary immunodeficiency

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study group: 100 children with suspicion of CD based on positive serology (TG2 >2 times upper limit of normal) and classical clinical manifestations or belonging to high risk groups, who underwent gastroscopy with intestinal biopsies.
  Control group: 100 children without suspicion of CD who underwent gastroscopy for other reasons (abdominal pain, failure to thrive, vomiting, eg)
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Celiac Disease based on histological findings. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Firas Rinawi, MD, Study Director — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider children's medical center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided